CLINICAL TRIAL: NCT04851730
Title: The Effect of an Individualized Impairment-based, Orthopedic Physical Therapy Intervention (IOI), on Muscle Stiffness, Pelvic Floor Function, and Pain in Women With Chronic Pelvic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Laurel Proulx, Principal Investigator, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FY2021-144
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Pain; Chronic Pain; Muscle Tightness
MeSH Terms: conditions — Pelvic Pain; Chronic Pain | interventions — Musculoskeletal Manipulations; Range of Motion, Articular; Exercise Therapy; Dry Needling

STUDY DESIGN:
Intervention Model Description: ABA single subject design
Masking Description: The researcher providing the orthopedic intervention will be blinded from the participant's pelvic floor muscle examination results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Orthopedic Intervention (Experimental): All subjects are receiving an orthopedic intervention that is specific to their presentation but made up of all intervention categories: Manual therapy, dry needling, deep breathing, stretching, strengthening, and progressive overload.
  Interventions: Procedure: Orthopedic Physical Therapy Intervention; Device: Dry Needling

INTERVENTIONS:
Procedure: Orthopedic Physical Therapy Intervention — First, a deep slow breathing protocol is intended to increase the expansion of the pelvic floor, utilizing the relationship between the diaphragm and the pelvic floor, resulting in a gentle stretching of the pelvic floor.
  Next, abdominal soft tissue mobilization, or scar mobilization of the lumbopelvic abdominal area will take place.
  Next, manual therapy to the thoracic or lumbar spine or the hips will be performed based on the impairments found in the orthopedic evaluation.
  The participant will be given a home exercise program to support breath training, and manual therapy. During the initiation of the second visit each participant will watch a standardized pain education video on the tablet, "Understanding pain in less than 5 minutes and what to do about it" The above plan of care will be completed 2 times/week for 4 weeks for a total of 8 visits.
  Other Names: manual therapy; mobility; deep breathing; graded exposure; therapeutic exercise
Device: Dry Needling — Third, the investigator will dry needle appropriate muscles. Dry needling treatment technique will include insertion of a sterile, disposable, solid filament needle into the muscle belly in the area palpated as listed below. A 0.30 × 0.50mm, or specified size below, stainless steel Seirin J-type or Myotech needle will be used (Dommerholt 2011). "Clean technique" will be employed throughout the treatment procedure which includes hand washing, clean latex-free glove use, and skin-surface preparation with an alcohol swab ( Baima & Isaac 2008). Each muscle will receive a maximal number of 2 insertions and each insertion consists of up to 5 seconds of a "pistoning" (in and out motion) technique in an attempt to elicit a local twitch response. Standard protocol for each muscle will be established prior to beginning data collection.
  Details about the dry needling protocol can be found in Appendix L.

SUMMARY:
The primary purpose of this study is to establish if an individualized, impairment-based orthopedic intervention (IOI) can improve pelvic floor function and pain in women with Chronic Pelvic Pain (CPP). Dry needling will be used as a part of the IOI to intervene upon peripheral muscles stiffness previously found to be more stiff in this population compared to healthy controls. This study is intended to initiate a line of research aimed at assessing widely used orthopedic physical therapy practices to address orthopedic impairments and muscle stiffness differences in women with CPP potentially decreasing time to care for a widely experienced condition. This study will guide potential future studies aimed at intervening upon a larger population and establishing the characteristics of participants who respond favorable to orthopedic care alone. First, this study will establish if this type of intervention has an effect on pelvic floor function and symptoms, pain, and muscle stiffness, all of which are often priorities of treatment for PHPTs treating CPP. A single-subject design is well suited in studying an intervention on such a heterogeneous patient population that does not currently have physical therapy treatment subclassifications. Future studies could help to establish possible subclassifications of CPP to include an orthopedic or peripheral muscle stiffness classification and empower therapists with associations between peripheral orthopedic and myofascial dysfunction and pelvic floor function and pain. This line of research could help prioritize which patients require specialty care, who could initiate care with an orthopedic PT, and who may resolve dysfunction and pain with orthopedic PT alone.

DETAILED DESCRIPTION:
When patients make their initial appointment at the private outpatient pelvic health office, they will be informed about a study looking for participants with pelvic pain that includes 4 weeks of free physical therapy care. If the patient is interested they will be given the researcher's email address and phone number to make appropriate arrangements. Once the potential participant contacts the researcher they will take part in a prescreening phone call. This prescreening call will assess their willingness to enroll in the study and ask preliminary inclusion criteria. This prescreening is necessary to allow participants to be taken off of the therapists' regular schedule and go onto the research schedule, allowing therapists to fill vacancies in their schedule if appropriate. If a participant emails or leaves a message, the researcher can call them to initiate the prescreening phone call. Potential subjects will be called a maximum of 2 times and up to 2 messages will be left for any potential subject that voiced interest by initiating contact with the researcher.

If the individual does not wish to participate after hearing more details from the researcher or for some reason does not meet inclusion criteria, the only information collected from the prescreening phone call will be gender, age, race, ethnicity, and reason for exclusion so that the number of patients that were screened compared to the number of patients that were enrolled, per the CONSORT guidelines, can be tracked. No further data will be collected or recorded from this call as it is intended to assess interest level and inform potential subjects that they will be scheduling with a researcher instead of a clinician. Individuals who contact researchers showing interest in the study from physician referral will also provide their contact information in order to schedule their first appointment with the researchers.

The information collected for prescreening or scheduling will only be shared with a small group of researchers in an encrypted file on a password protected computer. This file will be saved separately from any data collected by the study of enrolled participants. Enrolled subjects will be coded with a participant number as to not cross-identify with any record of contact information saved with the individual's name.

An ABA single-subject research design will be used for this study. Participants will undergo 3-5 sessions of baseline testing based on the stabilization of the dependent variable, with two visits per week until stabilization. If stabilization of two of the three dependent variables (NPRS, muscle stiffness, and PPT) can not be met then the participant cannot continue into the intervention phase of the study. Then the participants will undergo four weeks of intervention, two times a week for a total of 8 intervention appointments. Dependent variables will be collected one and two weeks after the last intervention ends to establish if there is a continuation of the data trend without intervention taking place.

15 women with CPP will be recruited as previously discussed. The participant will also be asked to wear a mask during the testing procedures and wash your hands before starting the session. First, we will take the participants temperature and ask if they have any symptoms of COVID-19, prior to each appointment. The researcher(s) will wash their hands with soap using methods recommended by the CDC before and after the research sessions. If hand washing is not available, we will use and ask them to use hand sanitizer. The researchers will also limit the number of research team members present to one treating member.

Unfortunately hands on intervention does not allow for social distancing. The researchers will conduct the study in a time efficient manner to minimize their time at the research site. The researcher(s) will wear masks during the entire study. If needed, the researchers will wear other PPE (personal protective equipment) such as laboratory coats or gowns, gloves, and eye protection during the study. When the researcher(s) must be in close proximity to the participants (e.g., performing the screening exam, performing manual therapy or dry needling), the researchers will have a face shield in addition to a mask.

After the participant has met inclusion and exclusion criteria and is enrolled in the study by Investigator #1, the participant will answer demographic and health history (Appendix A), pain, (Appendix B and C), psychosocial (Appendix F and G) and function and disability outcome measures (Appendix E). Next, Investigator #2 will perform a pelvic floor muscle assessment (Appendix D) in a private room at the consent of the participant and after informing the participant of the entire exam. Clean technique will be used with the therapist using one gloved finger with lubrication. The therapist will visually observe automatic and volition actions of shortening and lengthening of the pelvic floor and intra-vaginally manually assess the muscle strength of the superficial muscles consistent with the International Continence Society muscle grading system. Then the levator ani muscles will be assessed for power and endurance. All pelvic floor muscle measurements will be taken at each visit in the baseline and intervention phases, but will not be used as an outcome measure that determines stabilization.

Muscle stiffness measurements (Appendix C) will be collected using the MyotonPro by Investigator #1. MyotonPro measurements will be collected in the same order for each person to ensure similar resting time of each muscle. Testing will be done on the rectus femoris, adductor longus, lumbar paraspinals at levels L1/L2 and L4/L5 and the piriformis as these muscles were previously found to be significantly more stiff in those with CPP as compared to those without pelvic pain. Measurements of the individual muscles will be acquired on the more painful side if the participant is able to identify one, or by drawing a previously randomized card to determine the side of measurement. All measurements will be taken with the limb supported in a resting state. One measurement will be taken at each muscle due to previously acquired reliability measures. This measurement will establish if muscular stiffness is over 1 standard deviation (SD) above the average stiffness of a person without CPP, per muscle. If the person does have stiffness over 1SD, then dry needling will be performed on that muscle during the intervention phase of the study.

Next, PPT measurements (Appendix C) will be taken to assess local sensitivity to pain and pressure to measure changes in central sensitization over time at all muscle sites. PPT will also be assessed directly after dry needling is performed in the intervention phase. PPT measurements will be taken at all muscle sites, even if they do not meet the threshold to perform dry needling. A digital pressure algometer (Wagner Force Ten FDX, Wagner Instruments, Greenwich, CT) will be used to assess PPT. The algometer will be held by an examiner directly perpendicular to the muscle belly of and advanced at a rate of approximately 5N/sec. Participants will be instructed to verbally signal when they first perceive the force exerted as painful or uncomfortable.

After baseline measurements of pelvic floor muscle assessment, muscle stiffness, and PPT are complete, Investigator #1 will perform a standard lumbopelvic orthopedic exam (Appendix I). Based upon the preliminary MyotonPro testing and the orthopedic exam the intervention will be planned. This study is intended to replicate an individualized orthopedic plan of care using an impairment-based approach during the physical therapy evaluation. Since the intervention is based on what is found in the evaluation there is some discernment left up to the therapist. Standards will be established for each section of the orthopedic assessment in order to standardize which patient presentation gets what intervention as shown in Appendix J. The same order of care will be followed for each participant as well. Appendix J shows the possible interventions that can be performed based on each region of the evaluation. Documentation of the intervention and dosage will be recorded for each participant at each appointment.

The participants will be seen 2 times a week for 4 weeks for the intervention phase of the the A-B-A design.

Following the intervention portion of the study, the participant will come back for further dependent variable testing without intervention. The participant will return 1 time per week for 2 weeks. Measurements of PPT, muscle stiffness, NPRS, and pelvic floor and orthopedic function measurements will be taken at each visit through all phases of the study. Questionnaires such as the PFDI, CSI and BDI will be taken at the first baseline visit, last intervention visit and last follow-up visit since we do not expect these outcome measures to change from visit to visit.

ELIGIBILITY:
Inclusion Criteria:

* identified as female at birth and currently identifies as female
* between the ages of 18 and 50
* self identified pelvic pain for over 3 months and currently experiencing pain in the last week
* pain is non-cyclical in nature
* pain is located between the ilium, the umbilicus and pubic bone to include the vulva.

  * (Speer et al. 2016)

Exclusion Criteria:

* Participants will be excluded if they are experiencing pain due to reasons that are known to be inappropriate for orthopedic treatment such as acute fracture or malignancy, have a systemic condition which effects muscle stiffness measurements or meets a criteria that would change the validity or reliability of instrumentation, or have a medically serious reason for pelvic pain to include infection or neoplasm.

Exclusion criteria includes:

* body mass index >31(Bizzini & Mannion 2003)
* recent [3 month] history of pelvic surgery
* history of systemic inflammatory disease
* known pregnancy
* inability to lie prone, side and/or back for positioning of MyotonPro measurements or dry needling
* Inability to read and understand English
* current infection or neoplasm
* history of radiation therapy to any of the tissues being measured, (Lawrence et al. 2012)
* current fracture of lumbar spine, pelvis, hips or lower extremity
* received dry needling, injections, or soft-tissue mobilization of areas being measured within the past 4 weeks
* less than 6 months postpartum (Romano et al. 2010)

Additional exclusion criteria has been added due to the dry needling intervention. Exclusion criteria pertaining to dry needling includes:

* not giving consent to dry needling, having a needle phobia
* having a history of negative reaction to needling (or injection) in the past
* using anticoagulant therapy
* needling into an area or limb with lymphoedema as patients with lymphoedema may be more susceptible to infection
* abnormal bleeding tendency, thrombocytopenia,
* immunocompromised patients from disease (e.g. Blood borne disease, Cancer, HIV, AIDS, Hepatitis, bacterial endocarditis, incompetent heart valve or valve replacements etc.)
* immunocompromised from immunosuppression therapy or on cancer therapy
* acute immune disorders (E.G. acute states of rheumatoid arthritis, current infection, local or systemic etc.)
* has vascular Disease
* has epilepsy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — For the purposes of this study and to reduce the number of variables within the study that could contribute to pelvic pain, woman is defined as an individual who was identified as female at birth based on genitalia and currently identifies as female.
Enrollment: 15 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle stiffness pre- and post- dry needling and before and after the whole intervention | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks), immediately before and after dry needling (2 visits per week, weeks 2, 3, 4, 5 of the study)
  Using the MyotonPro peripheral muscles stiffness will be measures. Higher Nm equals more stiffness
Change in Pain Pressure Threshold, pre- and post- dry needling and before and after the whole intervention | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks), immediately before and after dry needling (2 visits per week, weeks 2, 3, 4, 5 of the study)
  Use a pressure algometer to test sensitivity to pressure. Less pressure equals more sensitivity.
Change in Numeric Pain Rating scale Pre- and Post- the whole orthopedic intervention | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks), immediately before and after dry needling (2 visits per week, weeks 2, 3, 4, 5 of the study)
  subjective outcome measure rating average pain through the week. Scale of 0-10 with 0 being no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Change in Subjective Pelvic floor muscle function Pre- and Post- the whole orthopedic intervention | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks)
  Pelvic floor distress inventory (PFDI-20). Scored on a scale of 0-100 with 100 being the maximum amount of distress a symptom causes

OTHER OUTCOMES:
Change in Pelvic Floor muscle function via intervaginal examination | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks)
  Intervaginal assessment of pelvic floor muscle strength rated on a scale of 0-5 with 5 being max strength and 0 being no contraction
Change in Pelvic Floor muscle function via intervaginal examination | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks)
  Intervaginal pelvic floor muscle endurance measured as the number of seconds they can hold the contraction up to 10 secs
Change in Pelvic Floor muscle function via intervaginal examination | difference between enrollment and end of intervention phase (5 weeks). Difference between end of intervention and end of follow-up (2 weeks)
  Intervaginal pelvic floor muscle coordination, being their ability to relax and bulge their pelvic floor volitionally

CONTACTS AND LOCATIONS:
Locations (1):
- Empower Your Pelvis, Lee's Summit, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baker PK. Musculoskeletal origins of chronic pelvic pain. Diagnosis and treatment. Obstet Gynecol Clin North Am. 1993 Dec;20(4):719-42. PMID 8115087
- [Result] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Result] Coronado RA, Bialosky JE. Manual physical therapy for chronic pain: the complex whole is greater than the sum of its parts. J Man Manip Ther. 2017 Jul;25(3):115-117. doi: 10.1080/10669817.2017.1309344. Epub 2017 Jun 12. No abstract available. PMID 28694673
- [Result] Dommerholt J. Dry needling - peripheral and central considerations. J Man Manip Ther. 2011 Nov;19(4):223-7. doi: 10.1179/106698111X13129729552065. PMID 23115475
- [Result] Jafari H, Courtois I, Van den Bergh O, Vlaeyen JWS, Van Diest I. Pain and respiration: a systematic review. Pain. 2017 Jun;158(6):995-1006. doi: 10.1097/j.pain.0000000000000865. PMID 28240995
- [Result] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648
- [Result] Loving S, Thomsen T, Jaszczak P, Nordling J. Pelvic floor muscle dysfunctions are prevalent in female chronic pelvic pain: a cross-sectional population-based study. Eur J Pain. 2014 Oct;18(9):1259-70. doi: 10.1002/j.1532-2149.2014.485.x. Epub 2014 Apr 3. PMID 24700500
- [Result] Maher RM, Hayes DM, Shinohara M. Quantification of dry needling and posture effects on myofascial trigger points using ultrasound shear-wave elastography. Arch Phys Med Rehabil. 2013 Nov;94(11):2146-50. doi: 10.1016/j.apmr.2013.04.021. Epub 2013 May 14. PMID 23684553
- [Result] Neville CE, Fitzgerald CM, Mallinson T, Badillo S, Hynes C, Tu F. A preliminary report of musculoskeletal dysfunction in female chronic pelvic pain: a blinded study of examination findings. J Bodyw Mov Ther. 2012 Jan;16(1):50-6. doi: 10.1016/j.jbmt.2011.06.002. Epub 2011 Jul 6. PMID 22196427
- [Derived] Proulx L, Brizzolara K, Thompson M, Wang-Price S, Rodriguez P, Koppenhaver S. Women with Chronic Pelvic Pain Demonstrate Increased Lumbopelvic Muscle Stiffness Compared to Asymptomatic Controls. J Womens Health (Larchmt). 2023 Feb;32(2):239-247. doi: 10.1089/jwh.2022.0198. Epub 2022 Nov 25. PMID 36450120